CLINICAL TRIAL: NCT05749588
Title: Precision Platform Study of Refractory Triple-negative Breast Cancer Based on Molecular Subtyping（(A Phase II, Open-label, Single-center Platform Study）
Brief Title: FUSCC Refractory TNBC Platform Study (FUTURE2.0)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N044
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Triple-negative Breast Cancer
Keywords: TNBC; Molecular Subtype; Precision Treatment; Platform Study
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- IM/HER2-low (Experimental): If patients were triple-negative breast cancer with IM subtype and HER2-low-positive
  Interventions: Drug: A1: SHR-A1811; Drug: A2: SHR-A1811 with Camrelizumab
- IM/HER2-0 (Experimental): If patients were triple-negative breast cancer with IM subtype and HER2-zero
  Interventions: Drug: B1: TROP2 ADC; Drug: B2: TROP2 ADC with Camrelizumab
- BLIS / HER2-low (Experimental): If patients were triple-negative breast cancer with BLIS subtype and HER2-low-positive
  Interventions: Drug: C1: SHR-A1811; Drug: C2: SHR-A1811 with BP102
- BLIS /HER2-0 (Experimental): If patients were triple-negative breast cancer with BLIS subtype and HER2-zero
  Interventions: Drug: D1: TROP2 ADC; Drug: D2: TROP2 ADC with BP102
- LAR / HER2-low (Experimental): If patients were triple-negative breast cancer with LAR subtype and HER2-low-positive
  Interventions: Drug: E1: SHR-A1811
- LAR /HER2-0 (Experimental): If patients were triple-negative breast cancer with LAR subtype and HER2-zero
  Interventions: Drug: F1: TROP2 ADC
- MES/ HER2-low (Experimental): If patients were triple-negative breast cancer with MES subtype and HER2-low-positive
  Interventions: Drug: G1: SHR-A1811
- MES /HER2-0 (Experimental): If patients were triple-negative breast cancer with MES subtype and HER2-zero
  Interventions: Drug: H1: TROP2 ADC

INTERVENTIONS:
Drug: A1: SHR-A1811 — A1: an anti-HER2 antibody-drug conjugate (ADC)
  Arms: IM/HER2-low
Drug: A2: SHR-A1811 with Camrelizumab — A2: SHR-A1811: an anti-HER2 antibody-drug conjugate (ADC)
  Camrelizumab: an anti-programmed death-1 (PD-1) antibody
  Other Names: SHR-1210
  Arms: IM/HER2-low
Drug: B1: TROP2 ADC — B1: an Trophoblast cell-surface antigen 2 (TROP2) ADC
  Arms: IM/HER2-0
Drug: B2: TROP2 ADC with Camrelizumab — B2: TROP2 ADC : an Trophoblast cell-surface antigen 2 (TROP2) ADC
  Camrelizumab: an anti-programmed death-1 (PD-1) antibody
  Other Names: SHR-1210
  Arms: IM/HER2-0
Drug: C1: SHR-A1811 — C1: an anti-HER2 antibody-drug conjugate (ADC)
  Arms: BLIS / HER2-low
Drug: C2: SHR-A1811 with BP102 — C2: SHR-A1811: an anti-HER2 antibody-drug conjugate (ADC)
  BP102: a humanized recombinant monoclonal IgG1 antibody (biosimilar to bevacizumab)
  Arms: BLIS / HER2-low
Drug: D1: TROP2 ADC — D1: an Trophoblast cell-surface antigen 2 (TROP2) ADC
  Arms: BLIS /HER2-0
Drug: D2: TROP2 ADC with BP102 — D2: TROP2 ADC : an Trophoblast cell-surface antigen 2 (TROP2) ADC
  BP102: a humanized recombinant monoclonal IgG1 antibody (biosimilar to bevacizumab)
  Arms: BLIS /HER2-0
Drug: E1: SHR-A1811 — E1: an anti-HER2 antibody-drug conjugate (ADC)
  Arms: LAR / HER2-low
Drug: F1: TROP2 ADC — F1: an Trophoblast cell-surface antigen 2 (TROP2) ADC
  Arms: LAR /HER2-0
Drug: G1: SHR-A1811 — G1: an anti-HER2 antibody-drug conjugate (ADC)
  Arms: MES/ HER2-low
Drug: H1: TROP2 ADC — H1: an Trophoblast cell-surface antigen 2 (TROP2) ADC
  Arms: MES /HER2-0

SUMMARY:
This is a Phase II, open-label, Single-center platform study research based on molecular subtypes to explore precision therapy in refractory triple-negative breast cancer.

DETAILED DESCRIPTION:
This is a Phase II, open-label, Single-center platform study，Based on FUSCC four TNBC subtypes and the results of the previous FUTURE trial, the investigators designed this platform trial, which for combined the TNBC subtyping and genomic sequencing-guided precision targeted therapy for refractory metastatic TNBC patients. In this trial, refractory mTNBC patients eligible for inclusion can be divided into various precision treatment group according to molecular typing and subtyping to evaluate the efficacy and safety of multiple precision targeted treatment. The research therapy arm can be updated with the update of basic translational research in our center, especially the refinement of typing, the discovery of new targets and the development of novel targeted drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥18 years;
2. TNBC invasive breast cancer confirmed by histology (specific definition: ER <1% positive tumor cells by immunohistochemistry are defined as ER negative, PR <1% positive tumor cells are defined as PR negative, HER2 0-1+ or HER2 ++ but negative by FISH without amplification was defined as HER2 negative); Locally advanced breast cancer (unable to undergo radical local treatment) or recurrent metastatic breast cancer;
3. Progression after at least one prior therapeutic regimens for advanced/metastatic TNBC
4. At least one measurable lesion according to RECIST 1.1 (conventional CT scan ≥20 mm, spiral CT scan ≥10 mm, measurable lesion has not received radiotherapy);
5. The functions of the main organs are basically normal and meet the following conditions:

   i. Blood routine examination criteria shall meet: HB ≥90 g/L (no blood transfusion within 14 days); The ANC acuity 1.5 x 10^9 /L; PLT acuity 75 x 10^9 /L;

   ii. Biochemical tests should meet the following criteria: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3×ULN; If liver metastases were present, ALT and AST≤ 5×ULN; Serum Cr ≤1×ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
6. They have not received radiotherapy, molecular targeted therapy, or surgery within 3 weeks before the start of the study, and have recovered from the acute toxicity of previous treatment (if surgery was performed, the wound has healed completely); No peripheral neuropathy or grade I peripheral neurotoxicity;
7. ECOG score ≤1, and life expectancy ≥3 months;
8. Fertile female subjects were required to use a medically approved contraceptive method during the study treatment period and for at least 3 months after the last use of the study drug;
9. Subjects volunteered to join the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Radiotherapy (except for palliative causes), chemotherapy, and immunotherapy were used in the first 3 weeks of treatment, except bisphosphonate (which can be used for bone metastasis);
2. Uncontrolled central nervous system metastases (indicating symptomatic or symptomatic treatment with glucocorticoids or mannitol);
3. A history of clinically important or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction, or ventricular arrhythmia within the last 6 months;
4. Persistent grade 1 or higher adverse reactions caused by previous treatments. The exception to this is hair loss or something the researchers don't think should be ruled out. Such cases should be clearly documented in the investigator's notes;
5. Underwent major surgery (except minor outpatient procedures, such as placement of vascular access) within 3 weeks of the first course of trial treatment;
6. Pregnant or lactating patients;
7. Malignancy (except basal cell carcinoma of the skin, which has been cured, and carcinoma in situ of the cervix) in the past 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study (approximately 3 years)
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study (approximately 3 years)
  Time to progressive disease (according to RECIST1.1)
Duration of Response (DoR) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study(approximately 3 years)
  Duration of whose best outcome is complete remission or partial remission (according to RECIST1.1)
Disease Control Rate (DCR) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study(approximately 3 years)
  The proportion of patients with the best overall response of CR, PR, or stable disease (SD)
Overall Survival (OS) | Randomization to death from any cause, through the end of study (approximately 3 years)
  Time to death due to any cause
CTCAE scale (V5.0) | Up to One Year during follow-up
  To evaluate the rate of adverse effects of patient by the standard CTCAE scale (V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No